CLINICAL TRIAL: NCT03952637
Title: A Phase 1/2 Study of Intravenous Gene Transfer With an AAV9 Vector Expressing Human Beta-galactosidase in Type I and Type II GM1 Gangliosidosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: Sio Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190101; 19-HG-0101
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12-09

CONDITIONS: Lysosomal Diseases; Gangliosidosis; GM1
Keywords: Lysosomal Diseases
MeSH Terms: conditions — Gangliosidoses | interventions — Rituximab; Sirolimus; Methylprednisolone; Prednisone; Absorptiometry, Photon; Electrocardiography; Echocardiography; Clinical Laboratory Techniques; Spinal Puncture; Catheterization, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 1 (Experimental): In Stage 1, up to 6 Type II subjects will receive 1.5E13 vg/kg of the gene transfer agent, up to 6 Type II subjects will receive 4.5E13 vg/kg, and up to 6 Type II subjects will receive 7.5E13 vg/kg of the gene transfer agent. In Stage 1, up to 3 Type I subjects will receive 1.5E13 of the gene transfer agent (Cohort 1) and up to 3 will then receive 4.5E13 of the gene transfer agent (Cohort 2).
  Interventions: Biological: AAV9-GLB1; Procedure: Abdominal ultrasound; Drug: Rituximab; Drug: Sirolimus; Drug: Methylprednisolone; Drug: Prednisone; Diagnostic Test: Audiology assessment with ABR; Diagnostic Test: Bone density scan (DEXA); Diagnostic Test: Electrocardiogram (EKG); Diagnostic Test: Echocardiogram; Other: Electroencephalogram (EEG) awake and extended overnight; Diagnostic Test: Laboratory tests; Procedure: Lumbar puncture; Procedure: Brain MRI/MRS/fMRI; Behavioral: Neurocognitive testing; Other: Neurology exam; Behavioral: PICC or other Central line placement; Procedure: Skeletal survey; Procedure: Skin biopsy; Procedure: Speech and modified barium swallow study; Procedure: Ophthalmology exam
- 2 (Experimental): Following the last Stage 1 subject s 6 months visit, data will be reviewed, and Stage 2 dosing and assessments will be determined. If Stage 2 dosing is to proceed, it will be reflected in a protocol amendment.
  Interventions: Biological: AAV9-GLB1; Procedure: Abdominal ultrasound; Drug: Rituximab; Drug: Sirolimus; Drug: Methylprednisolone; Drug: Prednisone; Diagnostic Test: Audiology assessment with ABR; Diagnostic Test: Bone density scan (DEXA); Diagnostic Test: Electrocardiogram (EKG); Diagnostic Test: Echocardiogram; Other: Electroencephalogram (EEG) awake and extended overnight; Diagnostic Test: Laboratory tests; Procedure: Lumbar puncture; Procedure: Brain MRI/MRS/fMRI; Behavioral: Neurocognitive testing; Other: Neurology exam; Behavioral: PICC or other Central line placement; Procedure: Skeletal survey; Procedure: Skin biopsy; Procedure: Speech and modified barium swallow study; Procedure: Ophthalmology exam

INTERVENTIONS:
Biological: AAV9-GLB1 — The risks of administering this treatment in a subject with GM1 gangliosidosis are not completely known. The major risk associated with intravenous infusion is from the subject s immunological response to the viral capsid and/or the beta-gal protein. To reduce this possibility, immune modulation therapy is being started prior to vector delivery and maintained for six months afterward. There is a theoretical risk that the integration of a small percentage of the rAAV vector DNA into the host cell genome could cause cellular transformation to cancer cells and lead to a malignancy. This has never been seen in subjects receiving intravenous AAV9 gene therapy so the risk of this complication, is likely very low.
Procedure: Abdominal ultrasound — Abdominal ultrasound will be performed as part of screening and safety follow- up studies. The ultrasound will be performed in a radiology department and will take approximately 20-30 minutes.
Drug: Rituximab — We are proposing the use of immune modulation to transiently deplete B-cells using rituximab. It will be infused at -21 days and -14 days before gene transfer.
Drug: Sirolimus — Sirolimus is a macrocytic lactone that inhibits T lymphocyte activation and proliferation by inhibiting activation of mammalian Target of Rapamycin (mTOR) kinase that suppresses cytokinedriven T-cell proliferation. We plan to give sirolimus from day -21 to Day 90 with option to extend to day 365 if clinically indicated.
Drug: Methylprednisolone — Subjects will receive IV methylprednisolone 1 mg/kg or a maximum dose of 50 mg, 60-120 minutes prior to vector administration on day 0 to mitigate potential acute innate immune response against the vector.
Drug: Prednisone — Prednisone (oral solution, dose 0.5 mg/kg) will be taken daily on Days 1-3.
Diagnostic Test: Audiology assessment with ABR — The audiology assessment will be performed in the Audiology Clinic using a standard audiogram to measure thresholds for pure tones and speech, word recognition, tympanometry, and otoacoustic emissions if the subject is capable and tolerant of these measures. The assessment will take approximately 30 minutes. The ABR is a noninvasive neurophysiologic test to evaluate electrical signal transmission from the 8th cranial nerve to the brainstem and the cortex in response to specific tones. Electrodes are placed on the scalp and on each earlobe. An earphone gives off a brief click or tone and the electrodes pick up the brain's responses to these sounds and record them. This will be performed by a trained neurophysiology technician to monitor possible change in hearing during treatment. The procedure will be performed in the Interventional Radiology suite while the subject is sedated following the MRI, fMRI, and MRS of the brain.
Diagnostic Test: Bone density scan (DEXA) — Type II subjects - This is a noninvasive enhanced form of X-ray that is used to measure bone loss. Loss of bone density is a known complication with GM1 gangliosidosis due to decrease in weight-bearing activities with disease progression. The procedure will be performed in the Nuclear Medicine Department. The subject s femur, spine, and whole body will be scanned at baseline and then yearly for 3 years. The procedure will take approximately 10 minutes and may be limited due to the subject s cooperation.
Diagnostic Test: Electrocardiogram (EKG) — Performed as part of screening and for safety before sedated procedures. The ECG will take approximately 10 minutes and may be limited due to the subject s cooperation.
Diagnostic Test: Echocardiogram — Performed as part of screening. The Echo will be done in the Echo Lab and may take approximately 20-30 minutes. The exam may be limited due to the subject s cooperation level.
Other: Electroencephalogram (EEG) awake and extended overnight — Completed at baseline. The subject will also have an EEG if clinically indicated (for example encephalopathy, seizures, or other change in neurological status or if changes on the previous study are deemed to warrant a follow up study) during post treatment follow up. The procedures will be conducted in the Neurology Testing Department. The total time for an awake EEG, including lead placement, is approximately 40 minutes. An extended overnight EEG will take approximately 12 hours. The exam may be limited due to the subject s cooperation level.
Diagnostic Test: Laboratory tests — Performed on blood and urine include safety labs, clinically indicated labs and research collections. Additional specimens may be collected for the PI s biorepository or as clinically indicated. Blood volumes for clinical diagnostic testing and research will be consistent with Clinical Center laboratory guidelines.
Procedure: Lumbar puncture — Performed to obtain cerebrospinal fluid (CSF) to measure GM1 ganglioside, beta-gal enzyme, AAV antibodies, Pentasaccharide biomarkers and other research tests. CSF will also be sent for cell count and differential, glucose, protein, and culture as well as CSF neurotransmitters. The amount of CSF obtained will be less than or equal to 0.75 mL/kg body weight. The procedure will be performed while under sedation following MRI imaging. If a sedated MRI is not being performed, then the LP will be performed in consultation with the pediatric consult service using conscious sedation and local anesthesia. The procedure will take approximately 15 minutes.
Procedure: Brain MRI/MRS/fMRI — Magnetic resonance imaging (MRI), functional MRI (fMRI) and spectroscopy (MRS) Procedure/Surgery - The subject will undergo noncontrast MRI, including DTI sequences, fMRI, and MRS in the 3T scanner using the same image acquisition sequences and the same MRS voxels to capture the same metabolites as prior sequencing under natural history protocol 02-HG0107. The MRI, fMRI, and MRS will be interpreted for signs of disease progression or stabilization and any signs of treatment toxicity by two board-certified radiologists with specialty training in neuroradiology. The scan will require anesthesia. Sedation will be administered by the anesthesia service after a preanesthesia consultation to assess risk. The type of sedation and whether the subject will be intubated for the procedure will be at the discretion of the anesthesia service.
Behavioral: Neurocognitive testing — Type II Subjects - The Vineland-3 will be administered under the supervision of a psychologist. The Vineland-3 provides several types of scores, measure of personal and social independence designed to examine the domains of communication, daily living skills, social skills and motor development. Other standard neurocognitive instruments may be used depending on the subject s ability, and some visits will (may) include a measure of intelligence /cognitive development if the child is able to achieve a basal score. Neurocognitive testing will take approximately 2-3 hours depending on subject cooperation. The assessments will not address sensitive topics. Type I Subjects - Bayley Scales of Infant and Toddler Development (BSID-III), a well-normed and validated, examiner-administered evaluation of cognition, language, and motor skills for children from birth to 42 months of age.
Other: Neurology exam — Neurology exam will be performed by a neurologist in the screening and followup appointments to monitor for any adverse reactions and to assess for clinical response to the treatment. The exam will be scripted for consistency within subject visits and between subjects and will take approximately 30 minutes to one hour. The exam will be videotaped. The exam may be limited due to the subject s cooperation level.
Behavioral: PICC or other Central line placement — PICC line or other central line placement will be done under sedation in Interventional Radiology. The procedure will be done under sedation and may take 20 minutes. A chest Xray will be done after placement to confirm correct positioning of the catheter.
Procedure: Skeletal survey — A skeletal survey will be performed to assess the degree of skeletal involvement of the disease. This will include X-rays of the a/p lateral spine, chest, and pelvis. The exam will take approximately 30 minutes. The exam may be limited due to the subject s cooperation level.
Procedure: Skin biopsy — Skin biopsy will be performed on subjects who have not already had a skin biopsy under the 02-HG-0107 protocol. The procedure will be done under sedation using local anesthetic. After washing the skin with chlorhexidine and numbing the skin with injectable lidocaine, a 3mm circle of skin is removed under sterile conditions and the wound is dressed. The entire procedure takes approximately 5 minutes.
Procedure: Speech and modified barium swallow study — Performed as a marker of response to treatment and safety. The swallow assessments will include a parental swallowing questionnaire and cranial nerve assessment. The NIH Swallowing Questionnaire from the Speech Language Pathology Section is designed to identify the presence and or absence of functional swallowing dysfunction as perceived by the subject and or caregiver. This 4point scale assists with further identification of clinical/research assessments of oral pharyngeal swallowing function if indicated in the form of a modified barium swallow. In addition to swallow assessments, tape recording of speech will also be included with diadochokinetic tasks and sustained phonations as well as speech if able. Recordings will be stored on a shared drive accessible only by the study team. The assessment may take approximately 30 minutes to 1 hour.
Procedure: Ophthalmology exam — The ophthalmology exam will be performed by an ophthalmologist in the screening and follow-up appointments to support subtype diagnosis and assess efficacy. Pictures of bilateral macula will be taken and saved to a secure database. OCT will also be performed. These exams will only be administered to Type I subjects.

SUMMARY:
Background:

GM1 gangliosidosis is a disorder that destroys nerve cells. It is fatal. There is no treatment. People with GM1 are deficient in a certain enzyme. A gene therapy may help the body make this enzyme. This could improve GM1 symptoms.

Objective:

To test if a gene therapy helps Type I and Type II GM1 gangliosidosis symptoms.

Eligibility:

Type I subjects will be male and female >= 6 months <= 12 months of age at the time of full ICF signing.

Type II subjects will be male and female > 12 months old and < 12 years old at the time of full ICF signing.

Design:

Participants will be screened with their medical history and a phone survey.

Participants will stay at NIH for 8-10 weeks.

Participants will have baseline tests:

Blood, urine, and heart tests

Hearing tests

Ultrasound of abdomen

EEG: Sticky patches on the participant s head will measure brain function.

Lumbar puncture: A needle will be stuck into the participant s spine to remove fluid.

MRI scans, bone x-rays, and bone scans: Participants will lie in a machine that takes pictures of the body

IQ tests

Neurology exams

Central line placement

Skin biopsy: A small piece of the participant s skin will be removed.

Speech tests

Participants will have an x-ray while swallowing food.

Participants will take drugs by mouth and IV. This will get their immune system ready for therapy.

Participants will get the gene therapy by IV. They may stay at NIH for a week to watch for side effects.

Participants will have visits 3 and 6 months after treatment. Then visits will be every 6 months for 2 years. Then they will have a visit at 3 years. Visits will take 4-5 days.

Participants will return to NIH once a year for 2 years for tests in an extension study....

DETAILED DESCRIPTION:
This is a non-randomized, Phase 1/2 clinical trial to study the safety and efficacy of a single dose gene transfer vector AAV9/GLB1 (AAV9-GLB1) by intravenous infusion to subjects with Type I and Type II GM1 gangliosidosis.

Type I subjects in this study will be male and female, >= 6 months old and <=12 months of age at the time of full ICF signing, with a diagnosis of Type I GM1 gangliosidosis. Type II subjects in this study will be male and female, > 6 months old and < 12 years old at the time of full ICF signing, with a diagnosis of Type II GM1 gangliosidosis. The subjects must have biallelic mutations in GLB1, a deficiency of Beta-galactosidase enzyme documented by testing in a CLIA-certified clinical laboratory, and serum AAV9 antibodies titers <= 1:50). Other inclusion/exclusion criteria apply. In Stage 1, up to 6 Type II subjects will receive 1.5E13 vg/kg of the gene transfer agent, and up to 6 Type II subjects will receive 4.5E13 vg/kg, and up to 6 Type II subjects will recieve 7.5E13 vg/kg of the gene transfer agent. In Stage 1, up to 3 Type I subjects will receive 1.5E13 of the gene transfer agent (Cohort 1) and up to 3 will then receive 4.5E13 of the gene transfer agent (Cohort 2). Dosing will be staggered to ensure subject safety.

Following the last Stage 1 subject s 6 months visit, data will be reviewed, and Stage 2 dosing will be determined. Up to 12 Type II and 6 Type I subjects are planned to be treated in Stage 2 of the study. If Stage 2 dosing is to proceed, it will be reflected in a protocol amendment.

The primary objective of Stage 1 of the study is to assess the safety of the AAV9-GLB1 vector following intravenous infusion. Stage 1 secondary and exploratory objectives include assessment of gene therapy on disease biomarkers, neurologic development and motor function, brain volume and myelination, and immune tolerance to the gene transfer vector.

Stage 2 of the study will assess the safety and efficacy of AAV9-GLB1 vector following intravenous infusion of the dose selected based on data from both Type I and II subjects.

Type I and Type II subjects have differing disease progression and symptomatology, justifying distinct endpoints and timepoint measures.

GM1 gangliosidosis is an autosomal recessive, neurodegenerative lysosomal storage disorder resulting from mutations in the GLB1 gene, encoding the enzyme Beta-galactosidase (Betagal). Betagal functions by removing terminal galactose moieties from GM1 ganglioside, a glycosphingolipid present in highest quantity in the CNS, primarily found in neurons. Betagal deficiency leads to accumulation of GM1 ganglioside and its asialo derivative (GA1) in the CNS. The age of onset and progression of GM1 gangliosidosis differs depending on the amount of residual Betagal activity, but the disease is generally divided into three clinical forms: Type I (infantile), Type IIa and IIb (late-infantile and juvenile), and Type III (adult or chronic). This clinical trial will treat GM1 Type I and Type II subjects.

The Type I form is the most severe, with age of onset less than 12 months of age and death often before age 3. Clinical findings of hypotonia and developmental delay/regression are found in almost all patients. In addition to symptoms resulting from severe CNS degeneration, evidenced by the presence of cherry-red maculae, infants often exhibit peripheral signs, including hepatosplenomegaly, skeletal dysplasia, cardiomyopathy, and coarse facial features.

The Type II form of GM1 generally has onset between 3 and 5 years with plateauing, then regression of developmental milestones (juvenile) or onset of symptoms after 12 months but before 24 months, plateauing of milestones then regression (late infantile).

Clinical features vary but in addition to CNS manifestations typically include a degree of skeletal involvement and mild hepatosplenomegaly. The primary symptoms are frequent falls, poor coordination, dysarthria and cognitive decline. Disease progression is variable, with subjects surviving well into the third decade (juvenile) or into the late teens (late infantile), but with severe cognitive and physical disabilities.

GM1 gangliosidosis is extremely rare, with an incidence estimated at 1:100,000 to 1:200,000. The disease is uniformly fatal with no effective therapy. Care is limited to symptomatic medical management. Intravenous administration of a gene transfer vector to deliver a normal copy of the GLB1 gene to the CNS could potentially provide an effective treatment for GM1 gangliosidosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Type I subjects

* Male or female subjects >= 6 months old and <= 12 months old at time of full ICF signing
* Biallelic mutations in GLB1
* Documented deficiency of Beta-galactosidase enzyme by clinical laboratory testing
* Phenotype consistent with a diagnosis of Type I GM1 gangliosidosis

  * Symptomatic subjects: as determined by the opinion of the Principal Investigator and based on the criteria set forth by Brunetti-Pierri et al:

    * Age of symptom onset <= 6 months of age
    * Rapidly progressive with developmental delay and hypotonia
  * Pre- symptomatic subjects: must have mutations confirmed to be associated with the Type I subtype
* AAV9 antibody titers <=1:50
* Agree to reside within 50 miles of the study site for at least 1 month following treatment

Type II subjects

* Vineland-3 Adaptive Behavior composite standard score greater than or equal to 40
* Male or female subjects > 6 months old and < 12 years old at time of full ICF signing
* Biallelic mutations in GLB1
* Documented deficiency of beta-galactosidase enzyme by clinical laboratory testing
* Phenotype consistent with a diagnosis of Type II GM1 gangliosidosis, with symptom onset after the first year of life
* AAV9 antibody titers <=1:50
* Agree to reside within 50 miles of the study site for at least 1 month following treatment

EXCLUSION CRITERIA:

* AAV9 antibody titers >1:50
* Contraindications to concomitant medications
* Serious illness that would not allow travel to the study site
* Unwilling to undergo study interventions as outlined in the Schedule of Events
* Subjects receiving other unapproved, off-label or experimental therapies for GM1 gangliosidosis (i.e. miglustat, Tanganil) within the last 60 days
* Any prior participation in a study in which a gene therapy vector or stem cell transplantation was administered
* Pregnant or lactating subjects
* Immunizations of any kind in the month prior to screening
* Evidence of cardiomyopathy on history, exam, or additional testing (echocardiogram or electrocardiogram) or other cardiac disease that in the opinion of the investigator would deem the subject unsafe to participate in the trial
* Indwelling ferromagnetic devices that would preclude MRI/fMRI/MRS imaging
* Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study
* History of infection with human immunodeficiency virus (HIV), hepatitis A, B, or C, or tuberculosis.
* History of or current chemotherapy, radiotherapy or other immunosuppressive therapy within the past 30 days. Corticosteroid treatment may be permitted at the discretion of the PI
* Abnormal laboratory values considered clinically significant per the investigator
* Failure to thrive, defined as:

  -- Falling 20 percentiles (20/100) in body weight in the 3 months preceding Screening/Baseline
* Underlying defect in immune function
* History of multiple and severe life-threatening infections

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Several time points over 3 years
  Assess the safety of the AAV9/GLB1 vector (AAV9-GLB1) following intravenous delivery.

SECONDARY OUTCOMES:
Brain MRI/MRS/fMRI | Varies between Type II and Type I subjects.
  Type II subjects - Assess brain volume using a 3T MRI, and central nervous system (CNS) metabolite levels by magnetic resonance spectroscopy (MRI) between pre- and post-treatment and compared to historical controls
CGI scale | Several timepoints over 3 years
  Type II subjects - Assess change in disease severity using the Clinical Global Impressions (CGI) scale.
Developmental changes | Varies between Type II and Type I subjects.
  Type II subjects: Assess developmental change in the Growth Scale Scores on the Vineland Adaptive Behavior Scales Third Edition (Vineland-3) instrument between pre- and post-treatment. Type I subjects - Bayley Scales of Infant and Toddler Development Third Edition (BSID-III) Composite score change from baseline
Motor function | Varies between Type II and Type I subjects.
  Type II subjects - Assess motor function using mobility scales developed as part of the natural history study
Neurological function | Several timepoints over 3 years
  Type I subjects - Neurological functional and developmental change from baseline
Overall survival | Throughout study
  Type I subjects life span is under 5 years
Diffusion tensor imaging | Comparing timepoints throughout the study. Varies between Type II and Type I subjects.
  Change in differential tractography using diffusion tensor imaging (DTI) pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Tifft, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
pending
Supporting Information: Study Protocol
Time Frame: pending
Access Criteria: pending

REFERENCES:
- [Derived] Lewis CJ, D'Souza P, Johnston JM, Acosta MT, Farmer C, Baker EH, Crowell A, Mojica Y, Ashraf S, Joseph L, Vezina G, Quezado Z, Yousef MH, Vardar Z, Shazeeb MS, Corti M, Blackwood M, Coleman K, Batista R, Thurm A, De Boever E, Gahl WA, Byrne BJ, Flotte TR, Jiang X, Gross AL, Keeler AM, Gray-Edwards H, Martin DR, Sena-Esteves M, Tifft CJ. AAV9 Gene Therapy in Type II GM1 Gangliosidosis - A Phase 1-2 Trial. N Engl J Med. 2026 Feb 6. doi: 10.1056/NEJMoa2510935. Online ahead of print. PMID 41665410
- [Derived] Lewis CJ, D'Souza P, Johnston JM, Acosta MT, Farmer C, Baker EH, Crowell A, Mojica Y, Rahman S, Joseph L, Hartman A, Vezina G, Quezado Z, Yousef MH, Luckett A, Vardar Z, Shazeeb MS, Corti M, Blackwood M, Coleman K, Thurm A, De Boever E, Gahl WA, Byrne BJ, Flotte TR, Jiang X, Gross AL, Keeler AM, Gray-Edwards H, Martin DR, Sena-Esteves M, Tifft CJ. AAV9 Gene Therapy in GM1 Gangliosidosis Type II: A Phase 1/2 Trial. medRxiv [Preprint]. 2025 Jul 29:2025.07.28.25332074. doi: 10.1101/2025.07.28.25332074. PMID 40766118
- [Derived] Liu S, Ma W, Feng Y, Zhang Y, Jia X, Tang C, Tang F, Wu X, Huang Y. AAV9-coGLB1 Improves Lysosomal Storage and Rescues Central Nervous System Inflammation in a Mutant Mouse Model of GM1 Gangliosidosis. Curr Gene Ther. 2022;22(4):352-365. doi: 10.2174/1566523222666220304092732. PMID 35249485
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-HG-0101.html